CLINICAL TRIAL: NCT00524992
Title: Prospective Evaluation of Albuminuria in HIV Positive Patients
Brief Title: Evaluation of Albuminuria HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070212; 07-DK-0212
Record Dates: First submitted 2007-09-01; First posted 2007-09-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-12-24

CONDITIONS: HIV-Associated Focal Segmental Glomerulosclerosis; HIV-Associated Collapsing Glomerulopathy; Proteinuria; Albuminuria; Renal Tubular Toxicity
Keywords: Focal Segmental Glomerulosclerosis; Collapsing Glomerulopathy; Anti-Retroviral Toxicity; Lipodystrophy; Metabolic Syndrome; Tubular Injury; Renal Biopsy; Proteinuria; Tenofovir Toxicity; HAART Toxicity; HIV Positive; HIV-Associated Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Proteinuria; Albuminuria; Glomerulosclerosis, Focal Segmental; Lipodystrophy; Metabolic Syndrome; HIV Seropositivity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the following: 1) how common albuminuria and proteinuria are among HIV-positive patients, 2) what causes albuminuria or proteinuria in these patients and 3) whether the condition becomes more severe over time. HIV-infected people are more likely than others to develop kidney disease. The earliest indicator of the possible presence of kidney disease is albuminuria (increased amounts of the protein albumin in the urine). A later indicator is the appearance of other proteins, a condition called proteinuria.

HIV-infected patients 8 years of age and older who do not have diabetes, chronic kidney disease or cancer may be eligible for this study.

Participants provide a urine sample during three visits as follows: the first upon enrollment in the study, a second 3 months later, and a third about 6 months after that. Blood samples are drawn at the first and last visits. At the first visit a medical history is taken and blood pressure, height, weight, waist circumference, hip circumference and upper arm skin thickness are measured.

Participants who are found to have albuminuria or proteinuria are asked to undergo a kidney biopsy for research purposes. The procedure is optional. Participants who develop heavy proteinuria may be recommended to undergo a kidney biopsy in order to determine the nature of the kidney disease and begin treatment. The biopsy requires a 2-day hospital stay. For the procedure, an anesthetic is given to numb the skin and a needle is inserted and guided into the kidney to withdraw a small tissue sample. The needle is passed twice, and possibly three times. Following the procedure, the subject remains in bed rest for at least 10 hours to minimize the risk of excessive bleeding.

DETAILED DESCRIPTION:
Problem: The appropriate approach to screening patients for early HIV-associated kidney disease is unknown. Recently, screening for microalbuminuria has been proposed; the clinical implications of finding microalbuminuria in this population are unknown, as several disease processes may contribute to microalbuminuria in this setting.

Background: Renal disease is becoming more common as patients with HIV disease live longer. Renal diseases in this population include glomerular diseases (collapsing glomerulopathy, immune complex glomerulonephritis, diabetic nephropathy, and hypertensive glomerulosclerosis) and various tubular diseases. Systemic endothelial dysfunction, occurring as part of metabolic syndrome and related disorders such as hypertension, hyperlipidemia, and insulin resistance, is also associated with microalbuminuria.

Study Objective: We wish to determine whether screening for microalbuminuria will detect early stage glomerular disease. We also wish to determine whether in some subjects renal histology is normal and microalbuminuria is a manifestation of metabolic syndrome, including HIV-associated lipodystrophy.

Design: We will use a cross-sectional study design.

Population: We will enroll 280 patients with HIV disease, to the extent practical enrolling consecutive patients in the NIAID Longitudinal HIV Clinic and the Washington Hospital Center HIV Clinic. This sample size was determined using an estimated population prevalence of microalbuminuria of 20%, with a 90% confidence interval of 5%. We will exclude patients with diabetes (as screening using urinary albumin excretion is well-established in clinical practice) and with established chronic kidney disease, defined as macroproteinuria (as these patients have been identified by a well-established screening test).

Methods: We will collect three urine samples, at three month intervals, for urine albumin/creatinine and protein/creatinine ratio. We will also collect data on blood pressure, anthropomorphometric parameters, and various serologic testing. Patients with persistent microalbuminuria will undergo renal biopsy. Using frozen blood cells, we will prepare DNA for genetic testing.

Analysis: We will determine the prevalence of microalbuminuria in the HIV population sample under study. We will determine the clinical implications of microalbuminuria, specifically how often HIV-associated collapsing glomerulopathy, HIV-associated glomerulonephritis, or other histologic disease is present. We will correlate the quantitative measure of urinary albumin with 1) the presence or absence of metabolic syndrome and with 2) various quantitative variables associated with metabolic syndrome. Finally, we will analyze kidney injury genes, in particular MYH9, to identify genes that predispose to microalbuminuria.

Future Studies: If this study suggests that the presence of microalbuminuria identifies patients who are likely to have early glomerular disease, we will consider undertaking a prospective controlled trial testing whether therapy with an angiotensin blocker can revert microalbuminuria and reduce progression to macroproteinuria.

ELIGIBILITY:
* INCLUSION CRITERIA:
* HIV+ adults and children greater than 8 years of age

EXCLUSION CRITERIA:

* Inability or unwillingness to give consent or assent or to comply with study requirements
* Unable to return to NIH or Washington Hospital Center for two follow-up visits over a 9-month period
* New opportunistic or bacterial infection within past 3 months or active opportunistic infection.
* Active malignancy, other than non-melanoma skin cancer and cutaneous Kaposi sarcoma not requiring treatment. Rationale: systemic inflammation may induce microalbuminuria.
* Diabetes by history
* IL-2, IL-7 or IFN-alpha therapy within past 3 months. Rationale: IL-2 and IFN-alpha therapy induce renal dysfunction and IL-7 may be associated with systemic inflammation.
* Non compliance, alcohol use, and drug use are conditions that make study completion unlikely or difficult.
* Diabetes (fasting glucose greater than 125 mg/dL or 2 hour oral glucose tolerance value greater than or equal to 200 mg/dL or current diagnosis of diabetes).
* Serum creatinine greater than 1.4 mg/dL.
* Urine protein/creatinine ratio greater than 0.5 and sustained on at least 2 measurements.
* Pregnant Women

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2007-08-29; Study Completion 2014-12-24

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Han TM, Naicker S, Ramdial PK, Assounga AG. A cross-sectional study of HIV-seropositive patients with varying degrees of proteinuria in South Africa. Kidney Int. 2006 Jun;69(12):2243-50. doi: 10.1038/sj.ki.5000339. Epub 2006 May 3. PMID 16672914
- [Background] Jones CA, Francis ME, Eberhardt MS, Chavers B, Coresh J, Engelgau M, Kusek JW, Byrd-Holt D, Narayan KM, Herman WH, Jones CP, Salive M, Agodoa LY. Microalbuminuria in the US population: third National Health and Nutrition Examination Survey. Am J Kidney Dis. 2002 Mar;39(3):445-59. doi: 10.1053/ajkd.2002.31388. PMID 11877563
- [Background] Chavers BM, Bilous RW, Ellis EN, Steffes MW, Mauer SM. Glomerular lesions and urinary albumin excretion in type I diabetes without overt proteinuria. N Engl J Med. 1989 Apr 13;320(15):966-70. doi: 10.1056/NEJM198904133201503. PMID 2784542
- [Derived] Hadigan C, Edwards E, Rosenberg A, Purdy JB, Fleischman E, Howard L, Mican JM, Sampath K, Oyalowo A, Johnson A, Adler A, Rehm C, Smith M, Lai L, Kopp JB. Microalbuminuria in HIV disease. Am J Nephrol. 2013;37(5):443-51. doi: 10.1159/000350384. Epub 2013 Apr 20. PMID 23615312